CLINICAL TRIAL: NCT07316192
Title: Outcomes With Pelashield™ PainGuard™ Compared to Restrata® in Standard Two-Stage Excision and Closure for Hidradenitis Suppurativa: A Prospective Cohort With Retrospective Comparator
Brief Title: Pelashield™ PainGuard™ vs Restrata® in HS Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Mark Granick, MD, FACS, MD, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2025001853
Record Dates: First submitted 2025-12-24; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Prospective; Wide local Excision; Wound Healing
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pelashield™ PainGuard™ Group (Experimental): Procedures:
  Perform wide excision of HS-affected tissue Apply Pelashield™ PainGuard™ to cover the surgical wound Place wound dressing and provide standard postoperative care instructions
  Interventions: Device: Pelashield Painguard

INTERVENTIONS:
Device: Pelashield Painguard — This is the only intervention being used in this study

SUMMARY:
Hidradenitis Suppurativa (HS) is a long-lasting skin condition that causes painful lumps and infections. In severe cases, patients need surgery to remove the affected skin. After surgery, a wound dressing called a wound matrix is placed over the area to help the skin heal.

This study will compare two different wound matrices:

Restrata®, which is the current standard treatment. Pelashield™ PainGuard™, a newer dressing that contains silver to reduce bacteria and lidocaine to help with pain.

The goal of this research is to find out if Pelashield™ PainGuard™ helps patients heal better after surgery than Restrata®. We will look at:

How quickly healthy granulation tissue (new healing tissue) forms How soon the wound is ready for the second surgery to apply a skin graft How often infections happen after surgery How much narcotic (opioid) pain medication patients need after surgery Patients who receive Pelashield™ PainGuard™ will be enrolled in the study going forward (prospective group). Patients who previously had surgery with Restrata® will be included through a review of their medical records (retrospective group). No additional procedures will be done outside of standard surgical care.

DETAILED DESCRIPTION:
Standard of Care vs. Research:

Wide surgical excision for Hidradenitis Suppurativa at University Hospital follows a standard two-stage approach: excision with wound matrix placement (Stage 1) followed by debridement and definitive closure with ReCell application (Stage 2). Currently, Restrata® wound matrix is our standard of care.

Research Component:

This study compares outcomes between our current standard (Restrata®) and an alternative FDA-cleared wound matrix (Pelashield™ PainGuard™) to determine whether Pelashield is a superior product. The research involves systematic data collection and comparison; all surgical procedures remain University Hospital standard of care.

Wide surgical excision for Hidradenitis Suppurativa following University Hospital's standard of care is often complicated by postoperative pain and poor skin graft adherence due to underlying bacterial overgrowth. Restrata® and Pelashield™ PainGuard™ are both synthetic wound matrices with FDA 510k clearance for use in surgical wounds. Pelashield™ PainGuard™ contains antimicrobial silver and local anesthetic, which may reduce postoperative pain and infection compared to Restrata®, and may provide a cleaner, more robust skin layer for enhanced wound healing and improved adherence of skin grafts. Additionally, the lower cost of Pelashield compared to Restrata aligns with University Hospital's commitment to responsible resource utilization and financial stewardship.

Specific Aim: To evaluate whether Pelashield™ PainGuard™, when used in place of Restrata® for wide excision of hidradenitis suppurativa, results in reduced narcotic pain medication use, reduced time to second procedure, and improved skin graft incorporation at wound site.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with a confirmed clinical diagnosis of HS requiring wide surgical excision.
* Ability to provide informed consent in English.
* Willingness and ability to attend routine postoperative follow-up visits to monitor healing and readiness for second-stage closure.

Exclusion Criteria:

* Non-English-speaking patients (due to consent and follow-up communication limitations).
* Known allergy or hypersensitivity to wound matrix components (polyvinyl alcohol), local anesthetics, or silver.
* Known sensitivity to lidocaine or history of cardiac conditions contraindicating lidocaine use (e.g., severe heart block, Adams-Stokes syndrome, Wolff-Parkinson-White syndrome).
* Pregnancy or active breastfeeding.
* Severe immunosuppression (e.g., chemotherapy within 3 months, solid organ transplant, uncontrolled HIV with CD4 <200, or chronic systemic steroids >10 mg prednisone-equivalent/day).
* Uncontrolled diabetes (most recent HbA1c >10% if available within 3 months).
* Active systemic infection or sepsis at time of surgery.
* Inability to complete postoperative follow-up through second-stage closure (e.g., plans to relocate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Postoperative Opioid Analgesic Usage | Period 1: After Stage 1 excision through day before Stage 2 closure (up to 8 weeks starting one day after surgery 1) Period 2: Stage 2 closure through 30 days post-Stage 2
  Total cumulative opioid consumption during two distinct postoperative periods:
ReCell Skin Graft Incorporation | Assessment performed at 14 days (±3 days) post-Stage 2 during routine clinic follow-up
  Percentage of the Stage 2 wound bed demonstrating successful ReCell graft take, reflecting the quality of granulation tissue and bacterial burden of the wound bed at time of grafting.
Surgical Site Infection (SSI) During Wound Bed Preparation | After Stage 1 excision through day before Stage 2 closure (up to 8 weeks starting one day after surgery 1)
  Presence of a clinically diagnosed surgical site infection occurring between Stage 1 excision and Stage 2 closure as defined by CDC criteria.
Time to Definitive Closure (Granulation Readiness) | After Stage 1 excision through day before Stage 2 closure (up to 8 weeks starting one day after surgery 1)
  Number of days from Stage 1 excision to Stage 2 definitive closure (debridement and ReCell application).

SECONDARY OUTCOMES:
Postoperative Non-Opioid Analgesic Use | Period 1: After Stage 1 excision through day before Stage 2 closure (up to 8 weeks starting one day after surgery 1) Period 2: Stage 2 closure through 30 days post-Stage 2

CONTACTS AND LOCATIONS:
Overall Officials: Mark Granick, MD, Principal Investigator — New Jersey Medical School
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
The findings from this study are intended to contribute to the scientific literature and will likely be disseminated through peer-reviewed publication or presentation at academic meetings. Participants will continue to receive all clinically relevant information about their own care and outcomes during routine follow-up visits, but they will not receive individual or aggregate research results unless they specifically request them after study completion.

REFERENCES:
- [Background] Leaper DJ, Schultz G, Carville K, Fletcher J, Swanson T, Drake R. Extending the TIME concept: what have we learned in the past 10 years?(*). Int Wound J. 2012 Dec;9 Suppl 2(Suppl 2):1-19. doi: 10.1111/j.1742-481X.2012.01097.x. PMID 23145905
- [Background] Wounds UK. International consensus. Appropriate use of silver dressings in wounds. Wounds UK. 2012;8(1):1-28.
- [Background] MacEwan MR, MacEwan S, Kovacs TR, Batts J. What Makes the Optimal Wound Healing Material? A Review of Current Science and Introduction of a Synthetic Nanofabricated Wound Care Scaffold. Cureus. 2017 Oct 2;9(10):e1736. doi: 10.7759/cureus.1736. PMID 29209583
- [Background] Matusiak L, Bieniek A, Szepietowski JC. Psychophysical aspects of hidradenitis suppurativa. Acta Derm Venereol. 2010 May;90(3):264-8. doi: 10.2340/00015555-0866. PMID 20526543
- [Background] Ring HC, Sorensen H, Miller IM, List EK, Saunte DM, Jemec GB. Pain in Hidradenitis Suppurativa: A Pilot Study. Acta Derm Venereol. 2016 May;96(4):554-6. doi: 10.2340/00015555-2308. No abstract available. PMID 26631388
- [Background] Scuderi N, Alfano C, Paolini G, et al. Surgical treatment of hidradenitis suppurativa: evaluation of two methods and postoperative outcome analysis. Int Wound J. 2013;10(4):435-441.
- [Background] Kohorst JJ, Baum CL, Otley CC, Roenigk RK, Schenck LA, Pemberton JH, Dozois EJ, Tran NV, Senchenkov A, Davis MD. Surgical Management of Hidradenitis Suppurativa: Outcomes of 590 Consecutive Patients. Dermatol Surg. 2016 Sep;42(9):1030-40. doi: 10.1097/DSS.0000000000000806. PMID 27340739
- [Background] Alavi A, Lynde C, Alhusayen R, Bourcier M, Delorme I, George R, Gooderham M, Gulliver W, Kalia S, Marcoux D, Poulin Y. Approach to the Management of Patients With Hidradenitis Suppurativa: A Consensus Document. J Cutan Med Surg. 2017 Nov/Dec;21(6):513-524. doi: 10.1177/1203475417716117. Epub 2017 Jun 22. PMID 28639459
- [Background] Mehdizadeh A, Hazen PG, Bechara FG, et al. A comprehensive review of surgical treatment in hidradenitis suppurativa. Dermatol Surg. 2015;41(Suppl 1):S149-S164.
- [Background] Jemec GB. Clinical practice. Hidradenitis suppurativa. N Engl J Med. 2012 Jan 12;366(2):158-64. doi: 10.1056/NEJMcp1014163. No abstract available. PMID 22236226